CLINICAL TRIAL: NCT03767062
Title: Comparison of Effects of Peripheral Nerve Block and Topiramate in the Treatment of Medication Overuse Headaches: A Randomised Parallel Group Study
Brief Title: Peripheral Nerve Block and Topiramate in the Treatment of Medication Overuse Headaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mustafa Ceylan, Principal İnvastigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/22-3
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Medication Overuse Headache; Chronic Migraine, Headache
Keywords: Medication overuse headache; Greater occipital nerve block; supratrochlear nerve block; topiramate.
MeSH Terms: conditions — Headache Disorders, Secondary; Headache | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topiramate (Active Comparator): Topiramate will be introduced 25 mg/day b.i.d. for the first week and increased to 100 mg/day b.i.d. for the second week.
  Interventions: Drug: Topamax
- Greater Occipital +Supratrochlear Nerve Block (Active Comparator): Greater occipital nerve block (GONB) will be applied to medial of the occipital artery which localized at the medial one-third of the superior nuchal line between the occipital tubercle and mastoid process. GONB solution is prepared with 1 ml triamcinolone (40mg), 2 ml bupivacaine (10 mg) and 1 ml 0,9% sodium chloride (NaCl). The injection is performed using a 22 gauge (G) × 1¼" (0.7 × 40mm) injector when the patient is lying prone on the table. The scalp is cleaned with iodine before procedure and injections are performed bilaterally with a volume of 2 mL after negative aspiration for blood. Supratrochlear nerve block (STNB) is applied 1 cm medial to superior orbital fissure using a mixture of 8 mg bupivacaine and 1.4 ml 0,9% NaCl. STNB is performed bilaterally with a volume of 1.5 mL after negative aspiration for blood.
  Interventions: Procedure: Greater Occipital Nerve Block + Supratrochlear Nerve Block

INTERVENTIONS:
Drug: Topamax — An antiepileptic agent used for migraine prophylaxis.
  Arms: Topiramate
Procedure: Greater Occipital Nerve Block + Supratrochlear Nerve Block — An injection to paralyze the occipital and supratrochlear nerves.
  Arms: Greater Occipital +Supratrochlear Nerve Block

SUMMARY:
Purpose: In this study, the investigators compared the effectiveness of peripheral nerve block (greater occipital nerve block with supratrochlear nerve block) versus topiramate as detoxification therapies in chronic migraine patients with medication overuse headache.

Methods: At least ninety chronic migraine patients with medication overuse headache are aimed to include in this study. Patients will be divided into the two groups. The first group will receive topiramate (n=45, estimated) and the second group will receive nerve block (n=45, estimated) as detoxification therapy. Patients' records regarding the visual analog scale (VAS) scores and headache frequencies are aimed to be collected before and after the therapy. Comparisons regarding VAS scores, headache frequencies, 50% responder rates and 75% responder rates will be performed in between topiramate and nerve block groups.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic migraine diagnosis according to International Classification of Headache-2 Disorders (ICHD)
2. w/o pregnancy or breastfeeding.
3. w/o acute or chronic psychiatric disorders.
4. w/o nephrolithiasis.
5. w/o medication of anticoagulant and antiaggregant.
6. w/o allergy to topiramate or bupivacaine.
7. w/o prophylaxis within the last three months with any of; propranolol, nebivolol, topiramate, valproate, venlafaxine, duloxetine, amitriptyline, flunarizine.
8. w/o previous history of peripheral nerve block, botulinum toxin or acupuncture.
9. w/o history of multiple sclerosis, movement disorders, epilepsy, stroke, and tumor.

J-w/o chronic systemic diseases including hypertension, cardiac insufficiency, diabetes, pulmonary disease, kidney disease, liver disease, and peripheral arterial disease.

Exclusion Criteria:

1. Lost to follow up within the pretreatment period during the detoxification therapy after the detoxification therapy
2. could not tolerate the peripheral nerve block or topiramate

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mustafa Ceylan, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zwart JA, Dyb G, Hagen K, Svebak S, Holmen J. Analgesic use: a predictor of chronic pain and medication overuse headache: the Head-HUNT Study. Neurology. 2003 Jul 22;61(2):160-4. doi: 10.1212/01.wnl.0000069924.69078.8d. PMID 12874392
- [Background] Grazzi L, Andrasik F, D'Amico D, Usai S, Kass S, Bussone G. Disability in chronic migraine patients with medication overuse: treatment effects at 1-year follow-up. Headache. 2004 Jul-Aug;44(7):678-83. doi: 10.1111/j.1526-4610.2004.04127.x. PMID 15209690
- [Background] Silberstein SD, Lipton RB, Dodick DW, Freitag FG, Ramadan N, Mathew N, Brandes JL, Bigal M, Saper J, Ascher S, Jordan DM, Greenberg SJ, Hulihan J; Topiramate Chronic Migraine Study Group. Efficacy and safety of topiramate for the treatment of chronic migraine: a randomized, double-blind, placebo-controlled trial. Headache. 2007 Feb;47(2):170-80. doi: 10.1111/j.1526-4610.2006.00684.x. PMID 17300356
- [Background] Tobin JA, Flitman SS. Occipital nerve blocks: effect of symptomatic medication: overuse and headache type on failure rate. Headache. 2009 Nov-Dec;49(10):1479-85. doi: 10.1111/j.1526-4610.2009.01549.x. PMID 19912347

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topiramate | Greater Occipital +Supratrochlear Nerve Block
Started | 45 | 45
Completed | 37 | 41
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate | Greater Occipital +Supratrochlear Nerve Block | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 45 | 90
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (7.1) | 32.9 (7.2) | 32.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 90
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 45 | 45 | 90
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale
Description: Range Pain 0-10, 0: No pain, 10: Worst Pain
Time Frame: Post treatment (4 weeks later)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Topiramate | Greater Occipital +Supratrochlear Nerve Block
Number analyzed (Participants) | 37 | 41
units on a scale
  Pretreatment (Baseline) | 8.3 (0.8) | 8.4 (0.7)
  Post treatment (4 weeks later) | 5.3 (1.2) | 5.3 (1.1)

2. Primary Outcome: Attack Frequencies
Description: Number of headaches patients suffer in a month.
Time Frame: Post treatment (4 weeks later)
Measure: Mean (Standard Deviation); unit: headaches per month
Arm/Group | Topiramate | Greater Occipital +Supratrochlear Nerve Block
Number analyzed (Participants) | 37 | 41
headaches per month
  Pretreatment (Baseline) | 21.2 (3.1) | 20.9 (2.7)
  Post treatment (4 weeks later) | 4.7 (2.8) | 5.9 (2.9)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Topiramate | Greater Occipital +Supratrochlear Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 2/45 | 0/45
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=45) | Greater Occipital +Supratrochlear Nerve Block (N=45)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) — Dizziness that affect concentration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-07): https://cdn.clinicaltrials.gov/large-docs/62/NCT03767062/Prot_SAP_000.pdf